CLINICAL TRIAL: NCT06516380
Title: Comprehensive Analysis of Cyberdyne HAL Single Joint, TecnoBody D-Wall, and Walker View 3.0 SCX Combined Therapy on Gait and Balance in a Post-Cartilage Knee Mosaicplasty Patient: A Detailed Case Study
Brief Title: Cyberdyne HAL, TecnoBody D-Wall, and Walker View 3.0 SCX Combined Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-45
Record Dates: First submitted 2024-07-04; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Mosaicplasty; Cyberdyne; Single Joint; TecnoBody

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- lower extremity strength (No Intervention): A 30 s sit and stand test was performed to evaluate lower extremity strength.
- walking test (No Intervention): The 10-metre walking test (10 MWT) and timed up and walk test (TUG) were performed.
- ROM (Experimental): Hip ROM, knee ROM, trunk flexion ROM were measured with TecnoBody Walker View 3.0 SCX device.
  Interventions: Device: Combined treatment of Cyberdyne HAL single joint with TecnoBody D-Wall and Walker View 3.0 SCX devices

INTERVENTIONS:
Device: Combined treatment of Cyberdyne HAL single joint with TecnoBody D-Wall and Walker View 3.0 SCX devices — HAL-SJ sessions were conducted 5 days a week for 3 months and 2 hours a day for a total of 60 sessions. HAL-SJ application was performed in cybernic voluntary control (CVC) mode for 90 minutes. In addition to each HAL-SJ session, balance exercises were performed with TecnoBody D-Wall for 30 minutes net.
  Arms: ROM

SUMMARY:
Mosaicplasty is a procedure where grafts taken from almost non-load-bearing areas of the joint are used to reconstruct lesioned areas. Hangody and his team developed this method using small cylindrical grafts and named it mosaicplasty (1). With the adoption of this approach, both the morbidity of the donor area has decreased, and a better joint surface has been achieved in the grafted area. Some studies have shown that 80% of this newly formed composite cartilage has a hyaline structure (2).

The Cyberdyne Hybrid Assistive Limb (HAL) - Single Joint (SJ) (HAL-SJ, Cyberdyne Inc., Tsukuba, Japan) is a wearable exoskeleton that facilitates voluntary control of knee joint movement. This exoskeleton processes signals from muscle action potentials detected by electrodes on the skin surface and assists the patient with joint movements. The knee joint power unit includes angular sensors and actuators, and the control system consists of Cybernetic Voluntary Control (CVC) and Cybernetic Autonomous Control (CAC) systems (3). HAL has been found to be effective in the functional improvement of various mobility disorders (4-7).

The TecnoBody Walker View (Bergamo, Italy) is used to analyze asymmetries and changes in joint range of motion. It can also be used to provide gait training, supporting weights ranging from 20% to 80%, and offers a safe walking rehabilitation option. The TecnoBody D-Wall is an assessment and rehabilitation device designed to improve movement quality with auditory and visual feedback. This device evaluates individuals' balance in seconds/mm² with eyes open (EO) and eyes closed (EC) conditions (8).

Although studies to date have reported successful outcomes for acute or chronic mobility disorders, there is limited literature on the use of HAL-SJ for cartilage rehabilitation or related postoperative recovery. Therefore, this study aims to investigate the effects of a combined treatment protocol involving HAL-SJ-based knee extension and flexion exercises with TecnoBody D-Wall and Walker View devices on gait parameters and balance during the acute recovery phase following mosaicplasty cartilage surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male patient aged 33 years.
* Body weight of 70 kg and height of 180 cm.
* Underwent knee mosaicplasty surgery on the right knee in November 2023.
* Presence of postoperative complications, including affected gait, reduced range of motion (ROM) in the knee joint, and edema.
* Ability to participate in intensive rehabilitation sessions (5 days a week, 2 hours per day) for 3 months.

Exclusion Criteria:

* Patients with severe cardiovascular, pulmonary, or neurological disorders that could affect participation in the rehabilitation program.
* Presence of any other musculoskeletal conditions that could interfere with the study outcomes.
* Patients with uncontrolled metabolic disorders such as diabetes.
* Inability to follow the prescribed rehabilitation protocol due to personal or logistical reasons.
* Participation in any other physical therapy or rehabilitation program during the study period.

Ages: 33 Years to 33 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Range of Motion | 4 weeks
  trunk flexion, hip flexion and knee flexion ROMs were measured at the end of the 20th session
Lower limb strength | 4 weeks
  A 30 s sit and stand test was performed to evaluate lower extremity strength.
Balance assessment | 4 weeks
  Balance assessment was performed on D-Wall device
10 metre walking test (10 MWT) | 4 weeks
  The 10 Meter Walking Test (10 MWT) is used to evaluate walking performance

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Etlik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided